CLINICAL TRIAL: NCT02286544
Title: Effects of Oxygen Treatment on Mechanisms Involved in Ischemia-reperfusion Injury: A Single Center, Randomized, Controlled Pilot Study in Healthy Volunteers
Brief Title: Effects of Oxygen Treatment on Mechanisms Involved in Ischemia-reperfusion Injury: A Pilot Study in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Leif Svensson, MD, PHD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DNR-2014/252-31; 2014-002282-30 (EudraCT Number)
Record Dates: First submitted 2014-10-27; First posted 2014-11-10 (Estimated); Last update posted 2017-12-11 (Actual); Status verified 2017-12

CONDITIONS: Myocardial Infarction; Inflammation; Acute Coronary Syndrome (ACS); Reperfusion Injury
Keywords: Myocardial Infarction; Oxygen; Inflammation; Acute coronary syndrome (ACS); ST-segment elevation myocardial infarction (STEMI); Reperfusion injury (IR-injury); Biomarkers; Normoxemia; Salmonella typhi; Vaccine-induced inflammation; Soluble markers of apoptosis; Leukocyte subset distribution; Matrix metalloproteinase (MMP); Biological Markers
MeSH Terms: conditions — Myocardial Infarction; Inflammation; Acute Coronary Syndrome; Reperfusion Injury; ST Elevation Myocardial Infarction | interventions — Vi polysaccharide vaccine, typhoid; Oxygen; Atorvastatin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Salmonella typhi vaccine (Active Comparator): 0.5 mL Salmonella typhi vaccine
  Interventions: Biological: Salmonella typhi vaccine (Typhim Vi®)
- Salmonella typhi vaccine + oxygen (Experimental): 0.5 mL Salmonella typhi vaccine + 6l/min oxygen
  Interventions: Biological: Salmonella typhi vaccine (Typhim Vi®); Drug: Oxygen (Oxymask®)
- S. typhi vaccine + oxygen + Atorvastatin (Experimental): 0.5 mL Salmonella typhi vaccine + 6l/min oxygen + 80mg Atorvastatin
  Interventions: Biological: Salmonella typhi vaccine (Typhim Vi®); Drug: Oxygen (Oxymask®); Drug: Atorvastatin

INTERVENTIONS:
Biological: Salmonella typhi vaccine (Typhim Vi®) — A peripheral venous catheter will be inserted. This catheter will be used to collect blood sample during the study day. In addition, peripheral oxygen saturation will be measured by pulse oximetry. After baseline venous blood samples have been collected, all study participants will receive 0.5 mL of the Salmonella typhi vaccine as an intramuscular injection (Typhim Vi®, Sanofi Pasteur MSD, injection solution 25 microgram/0.5 mL) Venous blood samples will be collected at 3, 6 and 8 hours after baseline. After the 8-hour blood sampling, the peripheral venous catheter will be removed and the study day ended.
Drug: Oxygen (Oxymask®) — As in arm 1. Half an hour after vaccination is administered, oxygen treatment will be initiated at 6 L/min via Oxymask® and continued for 6 hours. During oxygen treatment peripheral oxygen saturation will be measured by pulsoximetry.
  Venous blood samples will be collected at 3, 6 and 8 hours after baseline. After the 8-hour blood sampling, the peripheral venous catheter will be removed and the study day ended.
  Arms: S. typhi vaccine + oxygen + Atorvastatin; Salmonella typhi vaccine + oxygen
Drug: Atorvastatin — As in arm 1. Half an hour after vaccination is administered, oxygen treatment will be initiated at 6 L/min via Oxymask® and continued for 6 hours. During oxygen treatment peripheral oxygen saturation will be measured by pulsoximetry. A single dose of Atorvastatin 80 mg will be given immediately prior to start of oxygen. Venous blood samples will be collected at 3, 6 and 8 hours after baseline. After the 8-hour blood sampling, the peripheral venous catheter will be removed and the study day ended.
  Other Names: Lipitor
  Arms: S. typhi vaccine + oxygen + Atorvastatin

SUMMARY:
Oxygen treatment is widely used in acutely ill patients. In particular, oxygen treatment is routinely used in acute coronary syndrome (ACS) patients with suspected acute myocardial infarction and variably recommended in ACS-guidelines, despite very limited data supporting a beneficial effect.

Immediate re-opening of the acutely occluded infarct-related bloodvessel via primary percutaneous coronary intervention (PCI) is the treatment of choice to limit ischemic injury in the setting of ST-elevation ACS (STE-ACS). However, the sudden re-initiation of blood flow achieved with primary PCI can give rise to further damage, so-called reperfusion injury. Ischemia and reperfusion associated myocardial injury (IR-injury) involves a wide range of pathological processes. Vascular leakage, activation of cell death programs, transcriptional reprogramming, no reflow phenomenon and innate and adaptive immune activation all contribute to tissue damage, thereby determining the infarct size. The effect of oxygen treatment on these pathological processes, on the extent of IR-injury and the final infarct size in STE-ACS patients has not previously been studied.

ACS is characterized by a systemic inflammation with typical elevations of soluble inflammatory markers as well as changes in white blood cells. The inflammatory reaction might be considered helpful in restoring myocardial tissue structure and function, but on the other hand it might worsen IR-injury by activating various pathological processes. In human experimental studies, Salmonella typhi vaccine has been used to create a standardized model of systemic inflammation and when administered to healthy volunteers the vaccination has not been associated with any adverse events.

In an ongoing register randomized multicentre clinical trial, the DETO2X (Determination of role of oxygen in suspected acute myocardial infarction) study, the effect of oxygen on morbidity and mortality in ACS patients is being investigated. In a substudy of the DETO2X-trial, the investigators have planned to evaluate the effect of oxygen treatment on IR-injury in STE-ACS as assessed by biomarkers reflecting various aspects of the pathological processes involved.

The presented study is an experimental pilot study performed in healthy volunteers with a Salmonella typhi vaccine-induced inflammation with the purpose of studying effects of oxygen treatment on biological systems involved in the pathogenesis of IR- injury.

DETAILED DESCRIPTION:
HYPOTHESIS The main hypothesis is that oxygen treatment can increase oxidative stress, systemic inflammation, markers of apoptosis, matrix metalloproteinases (MMPs) and their tissue inhibitor (TIMPs) in individuals subjected to endotoxin-induced inflammation. The investigators also hypothesize that pretreatment with statins can prevent this oxygen effect.

AIMS

* To evaluate whether oxygen treatment can increase oxidative stress in healthy volunteers subjected to vaccine-induced inflammation.
* To assess the effect of oxygen treatment on plasma levels of soluble markers of apoptosis, MMPs and TIMPs in healthy volunteers with vaccine-induced inflammation.
* To study the effect of oxygen treatment on systemic inflammatory activity and leukocyte subset distribution in healthy volunteers with vaccine-induced inflammation.
* To evaluate the effect of oxygen treatment on platelet aggregation in healthy volunteers with vaccine-induced inflammation.
* To determine whether a potential oxygen effect on these cellular- and biomarkers can be prevented by pretreatment with Atorvastatin.
* To serve as a pilot study and basis for power calculations for a future planned study: "Effects of oxygen treatment on biomarkers of reperfusion damage and infarct size in ST-elevation myocardial infarction patients undergoing primary PCI".

DESIGN The present study is an experimental randomized pilot study in healthy volunteers.

STUDY POPULATION The investigators intend to include 36 healthy male volunteers. Females will not be included, due to the potential risk of hazardous effects of Salmonella typhi vaccine and Atorvastatin to a fetus in case of pregnancy.

STUDY DESIGN

At the time of inclusion all study participants will be randomised into one of three intervention groups:

Group 1) Salmonella typhi vaccine Group 2) Salmonella typhi vaccine + oxygen treatment Group 3) Salmonella typhi vaccine + oxygen treatment + Atorvastatin At 8.00 am on study day a peripheral venous catheter will be inserted. This catheter will be used to collect blood sample during the study day. In addition, peripheral oxygen saturation will be measured by pulse oximetry. After baseline venous blood samples have been collected, all study participants will receive 0.5 mL of the Salmonella typhi vaccine as an intramuscular injection (Typhim Vi®, Sanofi Pasteur MSD, injection solution 25 microgram/0.5 mL).

Half an hour after vaccination is administered, oxygen treatment will be initiated (in group 2 and 3) at 6 L/min via Oxymask® and continued for 6 hours. During oxygen treatment peripheral oxygen saturation will be measured by pulsoximetry. In group 3, a single dose of Atorvastatin 80 mg will be given immediately prior to start of oxygen. Venous blood samples will be collected at 3, 6 and 8 hours after baseline. After the 8-hour blood sampling, the peripheral venous catheter will be removed and the study day ended.

An experienced registered nurse and a resident or specialist in Cardiology and Internal Medicine will be present during the entire study day taking care of all study interventions, collecting blood samples and register data into the case report form (CRF) including potential adverse events.

EFFICACY OUTCOMES

* To determine the effect of oxygen treatment on biomarkers of oxidative stress, apoptosis, matrix metalloproteinases, markers of inflammation and platelet aggregation in healthy volunteers with Salmonella typhi vaccine-induced inflammation.
* To compare levels of these cellular- and biomarkers over time during an 8-hour study day.

SUMMARY The presented study is an experimental randomized pilot study performed in healthy volunteers with a Salmonella typhi vaccine-induced inflammation with the purpose of studying to date unknown effects of oxygen treatment on biological systems involved in the pathogenesis of IR- injury. As part of the DETO2X trial series, this study aims to contribute essential knowledge to clarifying the role of oxygen in treatment of acute myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 years
* Male gender

Exclusion Criteria:

* Female gender
* Not willing to participate
* Not able to communicate or to understand study instructions
* Participation in another on-going trial
* Any chronic disease
* Any acute disease within 30 days of study inclusion
* Any regular or temporary medication within 15 days of study inclusion
* Current smokers

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Plasma concentration levels over time of biomarkers of oxidative stress, apoptosis, inflammation and platelet aggregation | Within 8hours from baseline
  Venous blood samples will be collected at 3, 6 and 8 hours after baseline and plasmaconcentration analyzed for Interleukin (IL)-6 [pg/mL], CRP [mg/L], Isoprostane [pg/mL], Soluble TNF receptor 1 [pg/mL], Soluble TNF receptor 2 [pg/mL], Soluble Fas [pg/mL], Soluble Fas ligand (pg/mL], MMP-2 [ng/mL], TIMP-2 [ng/mL], Soluble P-selectin [ng/mL], Platelet factor (PF)-4 [ng/mL], Beta-thromboglobulin [ng/mL].

CONTACTS AND LOCATIONS:
Overall Officials: Lennart Nilsson, MD, PHD, Principal Investigator — Department of Medical and Health Sciences, Linköping University, and Department of Cardiology, University Hospital, 58185 Linköping, Sweden
Locations (1):
- Linköping University Hospital, Linköping, Sweden

REFERENCES:
- [Background] Hofmann R, James SK, Svensson L, Witt N, Frick M, Lindahl B, Ostlund O, Ekelund U, Erlinge D, Herlitz J, Jernberg T. DETermination of the role of OXygen in suspected Acute Myocardial Infarction trial. Am Heart J. 2014 Mar;167(3):322-8. doi: 10.1016/j.ahj.2013.09.022. Epub 2013 Dec 19. PMID 24576515
- [Background] Cabello JB, Burls A, Emparanza JI, Bayliss S, Quinn T. Oxygen therapy for acute myocardial infarction. Cochrane Database Syst Rev. 2013 Aug 21;(8):CD007160. doi: 10.1002/14651858.CD007160.pub3. PMID 23963794
- [Background] Yellon DM, Hausenloy DJ. Myocardial reperfusion injury. N Engl J Med. 2007 Sep 13;357(11):1121-35. doi: 10.1056/NEJMra071667. No abstract available. PMID 17855673
- [Background] Ekstrom M, Eriksson P, Tornvall P. Vaccination, a human model of inflammation, activates systemic inflammation but does not trigger proinflammatory gene expression in adipose tissue. J Intern Med. 2008 Dec;264(6):613-7. doi: 10.1111/j.1365-2796.2008.01998.x. No abstract available. PMID 19017180
- [Background] Eltzschig HK, Eckle T. Ischemia and reperfusion--from mechanism to translation. Nat Med. 2011 Nov 7;17(11):1391-401. doi: 10.1038/nm.2507. PMID 22064429
- [Background] Shuvy M, Atar D, Gabriel Steg P, Halvorsen S, Jolly S, Yusuf S, Lotan C. Oxygen therapy in acute coronary syndrome: are the benefits worth the risk? Eur Heart J. 2013 Jun;34(22):1630-5. doi: 10.1093/eurheartj/eht110. Epub 2013 Apr 3. PMID 23554440
- [Background] Piper HM, Meuter K, Schafer C. Cellular mechanisms of ischemia-reperfusion injury. Ann Thorac Surg. 2003 Feb;75(2):S644-8. doi: 10.1016/s0003-4975(02)04686-6. PMID 12607706